CLINICAL TRIAL: NCT06991621
Title: Mechanisms and Design Framework Study of Gamified Education in Professional Identity Formation for Medical Undergraduates
Brief Title: The Effect of Situation Puzzle Games on Nursing Students' Death Anxiety and Meaning in Life
Acronym: SPGI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenna Qian, Doctoral Researcher, School of Nursing, China Medical University, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Situation puzzle games-2025; 2024-FC7 (Other Grant/Funding Number: School of Nursing, China Medical University)
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Death Anxiety
MeSH Terms: conditions — Necrophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Education (Experimental): Scenario-based puzzle game in group sessions
  Interventions: Other: Puzzle game
- Manual Education (Active Comparator): Standardized death education manual
  Interventions: Other: Manual Education

INTERVENTIONS:
Other: Puzzle game — Scenario-based puzzle game sessions (group format)
  Arms: Gamified Education
Other: Manual Education — Standardized death education manual distribution
  Arms: Manual Education

SUMMARY:
Goal of this interventional study

The purpose of this research is to investigate the effects of a scenario-based puzzle educational game on death anxiety and meaning in life among nursing students. It aims to answer the following key questions:

Can the scenario-based puzzle educational game enhance nursing students' sense of meaning in life?

Can the scenario-based puzzle educational game reduce death anxiety in nursing students?

What are nursing students' experiences and perceptions of this educational game?

Study design Researchers will compare the intervention group (participating in the game) with a control group (receiving death education manuals) to evaluate the effectiveness of the game-based intervention.

Participants will:

Be recruited through campus posters

Be randomly assigned to either the intervention or control group and complete baseline questionnaires

In the control group: Receive death education manuals twice weekly for 3 weeks

In the intervention group: Participate in group sessions (5 students per group) to play the scenario-based puzzle game twice weekly for 3 weeks

Complete follow-up questionnaires and participate in qualitative interviews regarding their experiences with manual-based education or the game intervention after the 3-week intervention period

ELIGIBILITY:
Inclusion Criteria:

* Third-year full-time undergraduate nursing students
* Completed clinical observation training but not yet entered clinical internship phase
* Aged ≥18 years
* Provide informed consent and voluntarily participate in the study

Exclusion Criteria:

* Participated in similar death education interventions within the past 3 months
* Diagnosed with severe mental or psychological disorders
* Currently on a leave of absence (academic or personal)

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Death Anxiety | Week 0, Week 3
  A 15-item self-report scale developed by psychologist Templer (1967/1970) measuring death-related distress.
  Dimensions: Affective (Items 1,3,10,13,14), Stress/Pain (Items 4,5,6,9,11), Time Awareness (Items 8,12), Cognitive (Items 2,7,15)
  Scoring: Dichotomous (Yes/No) with 9 forward-scored and 6 reverse-scored items (Items 2,3,5,6,7,16*). Total score range: 0-15 (higher = greater anxiety).
  Reliability: Test-retest reliability (3-week) = 0.83; KR-20 = 0.76 (original English version).
Meaning in Life | Week 0, Week 3
  A 10-item scale (Steger et al.) assessing two dimensions:
  Presence of Meaning (5 items): Perceived life purpose
  Search for Meaning (5 items): Active pursuit of meaning
  Scoring: 7-point Likert (1="Strongly Disagree" to 7="Strongly Agree"). Higher scores indicate stronger meaning.
  Reliability: Cronbach's α = 0.878 (total), 0.850 (Presence), 0.907 (Search)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No